CLINICAL TRIAL: NCT04064411
Title: A Randomized, Non-inferiority, Phase 3, Open-label, Multicenter Study to Evaluate the Efficacy and Safety of Abaloparatide-sMTS for the Treatment of Postmenopausal Women With Osteoporosis (the wearABLe Study)
Brief Title: Efficacy & Safety of Abaloparatide-Solid Microstructured Transdermal System in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radius Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BA058-05-021
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Osteoporosis; transdermal delivery; microneedle; solid microstructured transdermal system; abaloparatide-sMTS; patch; abaloparatide; fracture; bone loss; TYMLOS®
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Fractures, Bone; Bone Diseases, Metabolic | interventions — abaloparatide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- abaloparatide-SC (Active Comparator): Participants self-administered daily doses of abaloparatide 80 mcg SC for 12 months using a single-participant, multiple-use, prefilled injection pen that delivers 30 doses. Participants received a new injection pen every 30 days.
  Interventions: Combination Product: abaloparatide
- abaloparatide-sMTS (Experimental): Abaloparatide-sMTS 300 mcg applied to the thigh for 5 minutes once daily for 12 months.
  Interventions: Combination Product: abaloparatide solid microstructured transdermal system

INTERVENTIONS:
Combination Product: abaloparatide — Abaloparatide is a synthetic peptide that is a potent and selective activator of the parathyroid hormone 1 receptor signaling pathway.
  Other Names: TYMLOS®; BA058; abaloparatide-SC
  Arms: abaloparatide-SC
Combination Product: abaloparatide solid microstructured transdermal system — Abaloparatide-sMTS is a drug-device combination product consisting of the drug abaloparatide coated onto a sMTS array for transdermal administration of abaloparatide.
  Other Names: BA058; abaloparatide-transdermal
  Arms: abaloparatide-sMTS

SUMMARY:
A 12-month study to compare the efficacy and safety of abaloparatide-solid microstructured transdermal system (sMTS) with abaloparatide-subcutaneous (SC).

DETAILED DESCRIPTION:
This study aims to evaluate the non-inferiority of abaloparatide-sMTS 300 micrograms (mcg) compared to abaloparatide-SC 80 mcg based on lumbar spine bone mineral density (BMD) at 12 months and to evaluate the safety and tolerability of abaloparatide-sMTS in the treatment of postmenopausal women with osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy ambulatory female from 50 to 85 years of age (inclusive) with postmenopausal osteoporosis
* Participants who are 50 to 65 years old with BMD T-score ≤ -2.5 and > -5.0 at the lumbar spine or hip (femoral neck or total hip) by dual energy x-ray absorptiometry (DXA) and meet one of the following: 1) radiological evidence of 2 or more mild or one or more moderate lumbar or thoracic vertebral fractures or 2) history of fragility fracture to the forearm, humerus, sacrum, pelvis, hip, femur, or tibia within the past 5 years.
* Participants older than 65 years with BMD T score ≤ -2.0 and > -5.0 who meet the fracture criteria may be enrolled
* Participants older than 65 years with BMD T score ≤ -3.0 and > -5.0 at the lumbar spine or hip (femoral neck or total hip) by DXA
* Body mass index of 18.5 to 33 kilograms (kg)/square meters (m^2), inclusive
* serum calcium (albumin-corrected), parathyroid hormone (1-84), serum phosphorus, alkaline phosphatase, and thyroid stimulating hormone within the normal reference range
* Serum 25-hydroxyvitamin D values must be ≥ 20 nanograms (ng)/milliliters (mL)

Exclusion Criteria:

* History of more than 4 mild or moderate spine fractures or any severe fracture
* Abnormality of the spine or hip that would prohibit assessment of BMD
* History of bone disorders other than postmenopausal osteoporosis or a diagnosis of cancer within the last 5 years
* History of Cushing's disease, thyroid, parathyroid, or malabsorptive syndromes or any chronic or recurrent diseases or disturbances that would interfere with the interpretation of study data or compromise the safety of the patient
* Prior treatment with parathyroid hormone, parathyroid hormone-related peptide-derived drugs, or bone anabolic steroids, including abaloparatide, teriparatide, or parathyroid hormone (1-84)
* Prior treatment with intravenous (IV) bisphosphonates at any time or oral bisphosphonates within the past 3 years; fluoride or strontium within the past 5 years; treatment with corticosteroids within the past 12 months; or selective estrogen receptor modulators within the past 6 months (except hormone replacement therapy)
* Prior treatment with an investigational drug or device within the past 90 days or 5 half-lives of the investigational drug, whichever is longer
* History of nephrolithiasis or urolithiasis within the past 5 years or hereditary disorders predisposing to osteosarcoma

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2021-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (97):
- United States (77):
  - University of Alabama Hospital at Birmingham, Birmingham, Alabama
  - Orthopedic Physician Alaska - Rheumatology, Anchorage, Alaska
  - Arizona Arthritis & Rheumatology Research, PLLC - Research Center - Glendale, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - SunValley Arthritis Center Ltd., Peoria, Arizona
  - Clinical Research Consortium, Tempe, Arizona
  - Arthritis & Rheumatism, Jonesboro, Arkansas
  - Advanced Clinical Research (ACR) - Rancho Paseo, Banning, California
  - Osteoporosis Medical Center, Beverly Hills, California
  - Clinical Trials of St. Jude Heritage Medical Group through S, Fullerton, California
  - Allied Clinical Research, Gold River, California
  - Marin Endocrine Care & Research, Inc., Greenbrae, California
  - St. Joseph Heritage Healthcare, Mission Viejo, California
  - Northern California Institute for Bone Health Inc., Orinda, California
  - Alta California Medical Group, Inc., Simi Valley, California
  - Lynn Institute of Denver, Aurora, Colorado
  - MedStar Georgetown University Hospital - Department of Obstetrics and Gynecology, Washington D.C., District of Columbia
  - UNC School of Medicine, Boca Raton, Florida
  - Bay Area Arthritis And Osteoporosis, Brandon, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Shrock Orthopaedic Research, LLC, Fort Lauderdale, Florida
  - Clinical Physiology Associates, an AMR company, Fort Myers, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - Health Awareness INC, Jupiter, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Rheumatic Wellness Institute, Miami, Florida
  - BDA Research, Miami, Florida
  - Center for Arthritis and Rheumatic Diseases, Miami, Florida
  - Sweet Hope Research Specialty, Miami Beach, Florida
  - Lakes Research, LLC, Miami Lakes, Florida
  - Global Health Research Center, Miami Lakes, Florida
  - Renstar Medical Research, Ocala, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Integral Rheumatology & Immunology Specialist, Plantation, Florida
  - Health Awareness, Inc., Port Saint Lucie, Florida
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Advanced Clinical Research (ACR) - Family Practice/General Medicine - Meridian, Boise, Idaho
  - St. Luke's Clinic - Rheumatology, Boise, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - MediSphere Medical Research Center, Evansville, Indiana
  - Northeast Iowa Medical Education Foundation, Waterloo, Iowa
  - Premier Medical Group, PSC, Owensboro, Kentucky
  - MedStar Health Center, Baltimore, Maryland
  - Rheumatology Consultants, Cumberland, Maryland
  - Othopaedic Associates of Michigan PC, Grand Rapids, Michigan
  - Montana Medical Research, Inc, Missoula, Montana
  - New Mexico Clinical Research, Albuquerque, New Mexico
  - The Endocrine Group, Albany, New York
  - Long Island Regional Arthritis & Osteoporosis Care PC, Babylon, New York
  - Physicians East, PA, Greenville, North Carolina
  - Cape Fear Arthritis Care, Leland, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Clinical Radiology Of Oklahoma, Edmond, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Dr. James Webb & Associates, Tulsa, Oklahoma
  - Altoona Center for Clinical Research - Research, Duncansville, Pennsylvania
  - PA Regional Center for Arthritis & Osteoporosis Research, Wyomissing, Pennsylvania
  - Palmetto Clinical Research, Summerville, South Carolina
  - The Endocrine Clinic PC, Memphis, Tennessee
  - Inquest Clinical Research, Baytown, Texas
  - Advanced Clinical Research-Be Well MD, Cedar Park, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Valley Institute of Research - General Practice, Harlingen, Texas
  - Valley Institute of Research, Harlingen, Texas
  - Biopharma Informatic LLC, Houston, Texas
  - Quality Research Inc., San Antonio, Texas
  - BFHC Research, San Antonio, Texas
  - Advanced Clinical Research (ACR) - Jordan Valley, West Jordan, Utah
  - Endocrinology & Diabetes Center, Chesapeake, Virginia
  - Western Branch Center for Women, Chesapeake, Virginia
  - Puget Sound Osteoporosis Center, Renton, Washington
  - Seattle Rheumatology Associates, Seattle, Washington
  - Arthritis Northwest Rheumatology, PLLC, Spokane, Washington
  - University of Wisconsin Madison, Madison, Wisconsin
- Denmark (3):
  - Center for Clinical and Basic Research A/S, Aalborg
  - Center for Clinical and Basic Research A/S, Ballerup Municipality
  - Center for Clinical and Basic Research A/S, Vejle
- Hungary (5):
  - Synexus Magyarország Egészségügyi Szolgáltató Kft. - Budapest, Budapest
  - Synexus Magyarország Egészségügyi Szolgáltató Kft. - Debrecen, Debrecen
  - Synexus Magyarország Egészségügyi Szolgáltató Kft. - Gyula, Gyula
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókórház, Nyíregyháza
  - Synexus Magyarország Egészségügyi Szolgáltató Kft. - Zalaegerszeg, Zalaegerszeg
- Poland (11):
  - Synexus Polska Sp. Z o.o. Oddział w Częstochowie, Częstochowa
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Specjalistyczny Osrodek Medycyny Wieku Dojrzałego Sp zo.o., Lodz
  - Synexus Polska Sp. Z o.o. Oddział w Lodzi, Lodz
  - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan
  - Specjalistyczny Ośrodek Medycyny Wieku Dojrzałego Sp. z o.o, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
- Mindful Rheumatix & Medical Research Group, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lewiecki EM, Czerwinski E, Recknor C, Strzelecka A, Valenzuela G, Lawrence M, Silverman S, Cardona J, Nattrass SM, Binkley N, Annett M, Pearman L, Mitlak B. Efficacy and Safety of Transdermal Abaloparatide in Postmenopausal Women with Osteoporosis: A Randomized Study. J Bone Miner Res. 2023 Oct;38(10):1404-1414. doi: 10.1002/jbmr.4877. Epub 2023 Jul 27. PMID 37417725

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible female participants were randomized to a 12-month open-label study treatment at 83 study centers in the United States, Denmark, Hungary, and Poland.
Groups:
- Abaloparatide-SC: Participants self-administered daily doses of abaloparatide 80 micrograms (mcg) subcutaneous (SC) using a single-participant, multiple-use, prefilled injection pen.
- Abaloparatide-sMTS: Participants self-administered daily doses of abaloparatide solid microstructured transdermal system (sMTS) 300 mcg.
Period: Overall Study
Arm/Group | Abaloparatide-SC | Abaloparatide-sMTS
Started (Intent-to-Treat (ITT) Population: Includes all participants randomized into this study.) | 255 | 256
Received at Least 1 Dose of Study Drug (Safety Population: Includes all participants who received at least 1 dose of study drug.) | 254 | 252
Completed | 191 | 201
Not Completed | 64 | 55
Not completed — Adverse Event | 29 | 19
Not completed — Significant Deterioration from Baseline (≥7%) of Bone Mineral Density (BMD) at Spine or Hip | 0 | 2
Not completed — Protocol Deviation | 0 | 2
Not completed — Withdrawal by Subject | 25 | 29
Not completed — Lost to Follow-up | 5 | 2
Not completed — Other than Specified | 4 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population (ITT): Includes all participants randomized into this study.
Groups:
- Abaloparatide-SC: Participants self-administered daily doses of abaloparatide 80 mcg SC using a single-participant, multiple-use, prefilled injection pen.
- Abaloparatide-sMTS: Participants self-administered daily doses of abaloparatide-sMTS 300 mcg.
- Total: Total of all reporting groups
Arm/Group | Abaloparatide-SC | Abaloparatide-sMTS | Total
Number analyzed (Participants) | 255 | 256 | 511
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (6.87) | 69.3 (6.49) | 69.1 (6.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 255 | 256 | 511
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 248 | 243 | 491
  Race: Black or African American | 4 | 4 | 8
  Race: Asian | 1 | 1 | 2
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Multiple | 0 | 3 | 3
  Race: Other | 2 | 4 | 6
  Ethnicity: Hispanic or Latino | 27 | 24 | 51
  Ethnicity: Not Hispanic or Latino | 227 | 230 | 457
  Ethnicity: Unknown | 1 | 2 | 3
Lumbar Spine BMD T-Score [Mean (Standard Deviation); unit: BMD T-Score] — The bone mineral density (BMD) T-score is the BMD, assessed by dual energy x-ray absorptiometry (DXA), at the site when compared to that of a healthy man/woman (20 to 29 years old). Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a man/woman (20 to 29 years old). Lower T-scores indicate worse bone condition. Population: Participants who had lumbar spine BMD T-Score assessment at baseline.
  BMD T-Score
    number analyzed (Participants) | 252 | 254 | 506
    (all) | -2.569 (1.1534) | -2.554 (1.0997) | -2.562 (1.1257)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 12
Description: Lumbar Spine BMD was assessed by DXA scans evaluated by a central imaging laboratory.
Time Frame: Baseline, Month 12
Population: Modified Intention-to-Treat (mITT): All randomized participants who received at least 1 dose of study drug and had a baseline lumbar spine BMD measurement and at least 1 postbaseline lumbar spine BMD measurement. Overall number of participants analyzed = participants with valid assessments at both baseline and Month 12.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Abaloparatide-SC | Abaloparatide-sMTS
Number analyzed (Participants) | 189 | 200
percent change | 10.8571 (0.4755) | 7.1361 (0.4605)
Statistical Analysis 1: Comparison: Abaloparatide-SC vs Abaloparatide-sMTS; Test type: Non-Inferiority — Noninferiority margin = 2.0% for abaloparatide-sMTS compared with abaloparatide-SC. Non-inferiority was to be concluded if the lower bound of the 2-sided 95% confidence interval (CI) for the estimated treatment difference (abaloparatide-sMTS minus abaloparatide-SC) in the percent change from baseline in lumbar spine BMD at 12 months was above -2.0% using a Mixed Model for Repeated Measures (MMRM) analysis; Least Squares Means (LSM) Difference = -3.7210, 95% CI 2-sided [-5.0089 to -2.4331] — LSM Difference = abaloparatide-sMTS minus abaloparatide-SC

2. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Month 12
Description: Total hip BMD was assessed by DXA scans evaluated by a central imaging laboratory.
Time Frame: Baseline, Month 12
Population: mITT: All randomized participants who received at least 1 dose of study drug and had a baseline lumbar spine BMD measurement and at least 1 postbaseline lumbar spine BMD measurement. Overall number of participants analyzed = participants with valid assessments at both baseline and Month 12.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Abaloparatide-SC | Abaloparatide-sMTS
Number analyzed (Participants) | 188 | 200
percent change | 3.6995 (0.2776) | 1.9688 (0.2675)

3. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD at Month 12
Description: Femoral neck BMD was assessed by DXA scans evaluated by a central imaging laboratory.
Time Frame: Baseline, Month 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Abaloparatide-SC | Abaloparatide-sMTS
Number analyzed (Participants) | 188 | 200
percent change | 3.4159 (0.3750) | 1.9163 (0.3599)

ADVERSE EVENTS:
Time Frame: Day 1 (after dosing) through Month 13
Description: All-Cause Mortality, Serious, and Other Adverse Events were assessed in the Safety Population: All randomized participants who received at least 1 dose of study drug.
Arm/Group | Abaloparatide-SC | Abaloparatide-sMTS
All-Cause Mortality (participants affected / at risk) | 1/254 | 0/252
Serious Adverse Events (participants affected / at risk) | 19/254 | 16/252
Other Adverse Events (participants affected / at risk) | 204/254 | 239/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abaloparatide-SC (N=254) | Abaloparatide-sMTS (N=252)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cannabinoid hyperemesis syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Normal pressure hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abaloparatide-SC (N=254) | Abaloparatide-sMTS (N=252)
Administration site erythema (General disorders) | 4 (4) | 13 (13)
Application site discolouration (General disorders) | 0 (0) | 37 (37)
Application site erythema (General disorders) | 15 (15) | 190 (205)
Application site haemorrhage (General disorders) | 2 (2) | 73 (78)
Application site oedema (General disorders) | 1 (1) | 122 (128)
Application site pain (General disorders) | 14 (23) | 142 (289)
Application site pruritus (General disorders) | 10 (10) | 83 (87)
Application site reaction (General disorders) | 0 (0) | 18 (20)
Application site swelling (General disorders) | 6 (6) | 116 (124)
Application site vesicles (General disorders) | 1 (1) | 16 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 (25) | 25 (29)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (34) | 14 (14)
COVID-19 (Infections and infestations) | 18 (18) | 9 (10)
Dizziness (Nervous system disorders) | 24 (28) | 17 (18)
Fatigue (General disorders) | 14 (14) | 6 (7)
Headache (Nervous system disorders) | 41 (46) | 25 (28)
Hypercalciuria (Renal and urinary disorders) | 6 (7) | 13 (13)
Hypertension (Vascular disorders) | 15 (16) | 8 (8)
Injection site bruising (General disorders) | 35 (37) | 1 (1)
Injection site erythema (General disorders) | 119 (131) | 26 (27)
Injection site haemorrhage (General disorders) | 30 (30) | 6 (6)
Injection site oedema (General disorders) | 31 (32) | 12 (12)
Injection site pain (General disorders) | 82 (164) | 17 (26)
Injection site pruritus (General disorders) | 48 (51) | 9 (9)
Injection site swelling (General disorders) | 48 (49) | 10 (10)
Nausea (Gastrointestinal disorders) | 35 (49) | 14 (14)
Orthostatic hypotension (Vascular disorders) | 20 (27) | 19 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (19) | 11 (15)
Palpitations (Cardiac disorders) | 18 (22) | 6 (7)
Urinary tract infection (Infections and infestations) | 20 (20) | 23 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04064411/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT04064411/SAP_001.pdf